CLINICAL TRIAL: NCT03728075
Title: The Role of Neuromuscular Electrical Stimulation in Regulation of Serum IL-6 and IL-15 in Chronic Heart Failure Patients
Brief Title: Neuromuscular Electrical Stimulation in Chronic Heart Failure Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 26/Panke.KKE/I/2017
Record Dates: First submitted 2018-10-24; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Chronic Heart Failure
Keywords: NMES; IL-6; IL-15; Chronic Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): standard protocol for cardiac rehabilitation
- Intervention group (Experimental): standard protocol for cardiac rehabilitation plus neuromuscular electrical stimulation (NMES)
  Interventions: Device: Neuromuscular electrical stimulation (NMES)

INTERVENTIONS:
Device: Neuromuscular electrical stimulation (NMES) — NMES was placed on the quadriceps muscle of both legs
  Arms: Intervention group

SUMMARY:
The purpose of the study is investigate the effects of NMES in regulation of serum IL-6 and IL-15 in chronic heart failure patients who received standard inpatient cardiac rehabilitation protocol

DETAILED DESCRIPTION:
Majority of chronic heart failure patients became intolerance of physical training that could limit activity. Recent studies reported that Neuromuscular electrical stimulation (NMES) application could increase muscle mass, oxidative enzyme, endothelial function, VO2 peak and quality of life in chronic heart failure patient. It was hypothesized that Neuromuscular Electrical Stimulation (NMES) assisted muscle contraction in chronic heart failure patients will increase the activity of myokine (Interleukin-6 and Interleukin-15), that in turn will promote exercise tolerance in this patient. the aim of this study was to investigate the effects of NMES in regulation of serum IL-6 and IL-15 in chronic heart failure patients who received standard inpatient cardiac rehabilitation protocol. Thirty chronic heart failure patients in cardiology ward that fulfilled inclusion criteria were randomized in two groups; the control group (standard inpatient cardiac rehabilitation protocol) and the intervention group (standard inpatient cardiac rehabilitation protocol and NMES). The intervention was done every day for seven days. Measurement of serum IL-6 and IL-15 were done before and after study, and analyzed by sandwich immunoassay with monoclonal antibody.

ELIGIBILITY:
Inclusion Criteria:

* heart failure patients admitted to the hospital NYHA II-III
* no weakness of lower limbs
* stable hemodynamic, already received standard treatment based on patient condition
* able to follow instruction
* lived at Surabaya or Sidoarjo
* assigned the informed consent

Exclusion Criteria:

* knee osteoarthritis with knee pain that interfere the ambulation
* phlebitis and active bleeding on lower limb
* use vasoactive drug (such as Dobutamin etc)
* already receive NMES before at femoris area in last 6 weeks before admission
* fracture of lower limb that interfere the ambulation
* sensory deficit at lower limb
* acute infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-21 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
IL-6 and IL-15 | before and 7th day of treatment
  pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Hening Laswati, Dr, Principal Investigator — Department of Physical Medicine and Rehabilitation, Faculty of Medicine Universitas Airlangga/ Dr Soetomo General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Faculty of Medicine Universitas Airlangga / Dr Soetomo General Hospital, Surabaya, East Java, Indonesia